CLINICAL TRIAL: NCT03878498
Title: Management of Anal Fistula of Crohn Disease
Acronym: FISTUCROHN
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC18_3041_FISTUCROHN
Record Dates: First submitted 2019-03-14; First posted 2019-03-18 (Actual); Last update posted 2019-03-18 (Actual); Status verified 2019-03

CONDITIONS: Anal Fistula; Crohn Disease
Keywords: Crohn disease; anal fistula; anal surgery
MeSH Terms: conditions — Rectal Fistula; Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: therapeutic management — therapeutic management of anal fistula in Crohn Disease

SUMMARY:
The management of anal fistula in Crohn Disease is complex. In aim to obtain the healing of the anal fistula, different approaches can be proposed but the best strategy is not yet determined. The aim was to describe the therapeutic management of anal fistula in Crohn Disease.

DETAILED DESCRIPTION:
Patients with anal fistula with Crohn disease and needed anal fistula drainage will be included. Medical and surgical treatments will be recorded. The management will be described and the best approaches will be identified.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age
* Crohn's disease with fistulizing anoperineal lesion
* Operated at least once for this reason

Exclusion Criteria:

* Adult person protected under the Public Health Code
* Minor person

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with anal fistula in Crohn Disease and needed fistula drainage or surgery
Sampling Method: Probability Sample
Enrollment: 212 (Estimated)
Dates: Start 2018-06-19 (Actual); Primary Completion 2019-09-19 (Estimated); Study Completion 2019-09-19 (Estimated)

PRIMARY OUTCOMES:
Description of the therapeutic management of anal fistula in Crohn Disease | The inclusion day
  Therapeutic management of anal fistula in Crohn Disease, including medical and surgical treatments

CONTACTS AND LOCATIONS:
Overall Officials: Charlène BROCHARD, MD, Principal Investigator — Rennes University Hospital
Locations (1):
- Centre Hospitalier Universitaire de Rennes, Rennes, France